CLINICAL TRIAL: NCT07378592
Title: Use Of Driving Simulator To Provide Pre-Driving Training For Adults With Acquired Brain Injuries.
Brief Title: Driving Simulator Training For Adults With Acquired Brain Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sacred Heart University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2025-237
Record Dates: First submitted 2026-01-15; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acquired Brain Injury
Keywords: Occupational Therapy; Pre-Driving; Behind-the-Wheel Assessments; Driving Simulation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving Simulator or Traditional Occupational Therapy as Pre-Driving intervention (Experimental): Participants will be randomly assigned to either the driving simulator (eight sessions) or eight sessions of traditional occupational therapy as a control group.
  Clients in the driving simulator intervention arm will receive eight sessions in a Drive Safety R-300 driving simulator. This simulator is a partial Ford Focus cab with a full interior, standard driving controls, and instrumentation, The exercises and realistic driving scenarios on the Drive Safety R-300 simulator will enable participants to have an immersive driving experience with interactive traffic, scripted behavior models, and triggered events. The researcher will initially provide more guided feedback during the motor tasks using a series of exercises in the simulator. More difficult motor tasks will be introduced gradually. As clients' motor skills became more refined, driving practice will be introduced in diverse scenarios and environmental conditions to improve the transfer and generalizability of motor skills.
  Interventions: Other: Driving Simulation Intervention
- Control - Traditonal Occupational Therapy (Active Comparator): Participants will be randomly assigned to either the driving simulator (eight sessions) or eight sessions of traditional occupational therapy as a control group.
  Participants in the control, occupational therapy group will receive interventions based on typical occupational therapy assessments which assess range of motion, strength, coordination, functional mobility and self care management. Participants will receive sessions that focus on their deficits using occupation-based interventions to improve their assessed deficits.
  Interventions: Other: Traditional Occupational Therapy

INTERVENTIONS:
Other: Driving Simulation Intervention — The exercises and realistic driving scenarios on the Drive Safety R-300 simulator will enable participants to have an immersive driving experience with interactive traffic, scripted behavior models, and triggered events. The researcher will initially provide more guided feedback during the motor tasks using a series of exercises in the simulator. More difficult motor tasks will be introduced gradually. As clients' motor skills became more refined, driving practice will be introduced in diverse scenarios and environmental conditions to improve the transfer and generalizability of motor skills.
  Arms: Driving Simulator or Traditional Occupational Therapy as Pre-Driving intervention
Other: Traditional Occupational Therapy — Traditional occupational therapy interventions are based on typical occupational therapy assessments which assess range of motion, strength, coordination, functional mobility and self care management. Participants will receive sessions that focus on their deficits based on their acquired brain injuries. The researcher will use occupation-based interventions to improve the participants performance in functional tasks and performance in areas of occupations such as self care, leisure, play, health care management, and work.
  Arms: Control - Traditonal Occupational Therapy

SUMMARY:
The aim of this project is to prepare adults with acquired brain injuries for on-road driving by using the driving simulator and increase participant's comfort level, confidence, and independence within their occupation of driving. The occupational therapy faculty are interested in identifying the impact driving simulation training has on individuals with acquired brain injuries and how it prepares them for on-road driving. We hope that the information from this project will help us gather information on how driving simulation training improves pre-driving skills related to comfort, confidence, and independence.

DETAILED DESCRIPTION:
This is Phase 3 of a project that started as a capstone project in 2021 and continued with Phase 2 in 2022. . In this next phase,participants who qualify for the study will be invited to participate in the study and will be sent a consent form. They will be randomly assigned to either the driving simulator (eightsessions) or eight sessions of traditional occupational therapy as a control group. All participants will have pre- and post-testing using the same assessments. These assessments measure readiness-to-drive. All participants in the control group will be offered drivingsimulator training after completing the traditional occupational therapy sessions. All study participants will be referred to a certified driving rehabilitation specialist for behind-the-wheelassessments after completing of the driving simulation training

ELIGIBILITY:
Inclusion Criteria:

* Adult participants over 18 years
* Diagnosed acquired brain injury
* A valid driver's license
* History of driving prior to injury

Exclusion Criteria:

* Age less than 18 years
* Moderate to severe cognitive impairment, as measured on the Montreal Cognitive Assessment
* Visual acuity or visual field issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Useful Field of View Assessment | 8-16 weeks
  This is a cognitive assessment that reliably predicts crash risk in drivers. There are 3 sub tests: Processing Speed, Divided Attention, and Selective Attention, which are measured in milliseconds (ms). The 3 sub-tests contribute to an Index score which ranges from 1-5 (Very Low Risk to High Risk of vehicular crash)
Motor Free Visual Perceptual Test | After 16 intervention sessions
  This assessment measure is meant to assess visual perception independent of motor ability. The unit of measurement is age equivalent in years and months
Trails A and B assessment | 8-16 weeks
  This are tests of speed for attention, sequencing, mental flexibility, visual search, and motor function. The subject is required to connect 25 encircled numbers by pencil line (Part A) and 25 alternating encircled numbers and letters (Part B) in correct order. The unit of measurement is seconds.

SECONDARY OUTCOMES:
Behind-the-Wheel Assessment | 8-16 weeks
  Participants will be referred to a certified driving rehabiliation specialist for a behind-the-wheel assessment after completing their 8 intervention sessions. The unit of measurement is Pass or Fail

CONTACTS AND LOCATIONS:
Overall Officials: Sheelagh Schlegel, DrHSc, MPH, OTR/L, Principal Investigator — Sacred Heart University
Locations (1):
- Sacred Heart University, Fairfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on the study protocol for the driving simulation and data showing performance on the neuropsychological assessments
Supporting Information: Study Protocol, CSR
Time Frame: 1/1/2027 - 12/31/2029
Access Criteria: Driving Simulation researchers

REFERENCES:
- [Background] Blane A, Lee HC, Falkmer T, Willstrand TD. Assessing Cognitive Ability and Simulator-Based Driving Performance in Poststroke Adults. Behav Neurol. 2017;2017:1378308. doi: 10.1155/2017/1378308. Epub 2017 May 7. PMID 28559646
- [Background] Dickerson AE, Meuel DB, Ridenour CD, Cooper K. Assessment tools predicting fitness to drive in older adults: a systematic review. Am J Occup Ther. 2014 Nov-Dec;68(6):670-80. doi: 10.5014/ajot.2014.011833. PMID 25397762
- [Background] Ouellette DS, Kaplan S, Rosario ER. Back on the Road: Comparing Cognitive Assessments to Driving Simulators in Moderate to Severe Traumatic Brain Injuries. Brain Sci. 2022 Dec 28;13(1):54. doi: 10.3390/brainsci13010054. PMID 36672036
- [Background] Frankish JG. Day hospital fees and accessibility of essential health services. S Afr Med J. 1986 Aug 30;70(5):285-8. PMID 3750125
- [Background] Dimech-Betancourt B, Ross PE, Ponsford JL, Charlton JL, Stolwyk RJ. The development of a simulator-based intervention to rehabilitate driving skills in people with acquired brain injury. Disabil Rehabil Assist Technol. 2021 Apr;16(3):289-300. doi: 10.1080/17483107.2019.1673835. Epub 2019 Oct 9. PMID 31597483

DOCUMENTS (1):
  • Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT07378592/ICF_000.pdf